CLINICAL TRIAL: NCT01991158
Title: An Open, Single-center, Phase II Clinical Trial for Treatment of Untreated Extranodal NK/T Cell Lymphoma With High Dose of Methotrexate in Combination With Gemcitabine, Pegaspargase and Dexamethasone (GAD-M Regimen)
Brief Title: GAD-M Regimen As First-Line Treatment in Untreated Extranodal NK/T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Li Zhiming, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2013-030-01
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Extranodal NK/T-cell Lymphoma, Nasal Type
Keywords: GAD-M regimen; first line chemotherapy; NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Methotrexate; Gemcitabine; pegaspargase; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GAD-M regimen (Experimental): GAD-M regimen means High dose of methotrexate combined with gemcitabine, pegaspargase and dexamethasone
  Interventions: Drug: High dose of methotrexate; Drug: Gemcitabine; Drug: Pegaspargase; Drug: Dexamethasone

INTERVENTIONS:
Drug: High dose of methotrexate — Methotrexate 3.0g/Kg, intravenous drip D1
Drug: Gemcitabine — Gemcitabine 1g/m2 intravenous drip D1,D8
Drug: Pegaspargase — Pegaspargase 2500U/m2 intramuscular injection (IM) D1
Drug: Dexamethasone — Dexamethasone 20mg/d intravenous drip D1, po D2-3

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of High dose of Methotrexate combined with gemcitabine, pegaspargase and dexamethasone (GAD-M regimen) as first-line treatment in patients with de novo extranodal NK/T cell lymphoma.

DETAILED DESCRIPTION:
Studies have shown that effects of P glycoprotein mediated chemotherapy resistance reduce the therapeutic efficacy of anthracycline-based chemotherapy of NK/T cell lymphoma, and agents like pegaspargase and large doses of Methotrexate is not affected by the P glycoprotein. A number of reports suggest that gemcitabine combined with other chemotherapy drugs has good application prospect in the treatment of lymphomas. Dexamethasone is used in combination with other agents for the treatment of lymphomas which may be implicated in the development or growth of some cancers. So we explored to evaluate the efficacy and safety of High dose of methotrexate combined with gemcitabine, pegaspargase and dexamethasone (GAD-M regimen) as first-line treatment in patients with untreated extranodal NK/T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of NK/T Cell Lymphoma;
* Age:18-80 years;
* Weight：Male：67±20Kg（47-87Kg），Female：55±20Kg（35-75Kg）
* Eastern Cooperative Oncology Group (ECOG) status 0-3, Estimated survival time > 3 months;
* No history of other malignancies; No other current tumors；
* Normal haematological, liver and renal function (WBC count≥3.5×109/L, Hemoglobin≥100g/L, platelet count≥90×109/L, bilirubin<1.5×ULN, Alanine transaminase (ALT) and Aspartate Aminotransferase (AST)<2.5×ULN, serum creatinine<1.5×ULN), normal coagulation function and cardiac function;
* Clinical staging I-IV；
* No previous treatments including chemotherapy, radiotherapy, targeted therapy or stem cell transplantation;
* Appreciable and measurable lesions, clinical assessment >2cm，CT or MRI >1.5cm;
* No other serious diseases which conflict with the treatment in the present trial;
* No concurrent treatments that conflict with the treatments in the present trial(including steroid drugs);
* Voluntary participation and signed the informed consent.

Exclusion Criteria:

* The patients had the conditions below: clinically significant ventricular tachycardia (VT), atrial fibrillation (AF), heart block, myocardial infarction (MI), congestive heart failure (CHF), symptomatic coronary artery heart disease requiring medication;
* The patients suffered from organ transplant
* The patients participated in other clinical trials within the 30 days before enrollment or who are participating in other clinical studies;
* The patients with active bleeding or new thrombotic disease, who are taking anticoagulant drugs or with a history of bleeding tendencies，who with active infection;
* The patients suffered before surgery less than four weeks, or after less than six weeks;
* The patients with abnormal liver function (total bilirubin> 1.5 times the normal value, ALT / AST> 2.5 times normal), abnormal renal function (serum creatinine> 1.5 times normal), blood abnormalities (absolute neutrophil count <1.5 × 109 / L, platelets <80 × 109 / L, hemoglobin <90g /L) ;
* The patients with mentally ill / unable to obtain informed consent;
* The patients with drug addiction, alcohol abuse which affects the long-term evaluation of test results;
* The patients in pregnancy, lactation and women of childbearing age who do not want to take contraceptive measures subjects;
* Clinical and laboratory support brain metastases;
* The patients with a history of allergy or adverse reaction(s) to test drug;
* The patients not suitable to participate in the investigator judged by researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-12 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | every 6 weeks, up to completion of treatment (approximately 6 months)
  21 days (3 weeks) for one cycle, Efficacy was evaluated every two cycles

SECONDARY OUTCOMES:
Progress Free Survival (PFS) | up to end of follow-up-phase (approximately 5 years)
Overall Survival (OS) | up to the date of death (approximately 5 years)

OTHER OUTCOMES:
The number of participants with adverse events of grade 3-4 | every 3 weeks, up to completion of treatment (approximately 6 months)
  21 days (3 weeks) for one cycle, Toxicity was evaluated every cycle
Epstein-Barr virus(EBV) DNA copies and antibodies | every 3 weeks,up to completion of treatment(approximately 6 months)
  21 days(3 weeks) for one cycle
Plasma β2-microglobulin | every 3 weeks,up to completion of treatment(approximately 6 months)
  21 days(3 weeks) for one cycle
Urinary microglobulin β2 | every 3 weeks,up to completion of treatment(approximately 6 months)
  21 days(3 weeks) for one cycle
lymphocyte count | every 3 weeks,up to completion of treatment(approximately 6 months) 21
  21 days(3 weeks) for one cycle
Monocyte Count | every 3 weeks,up to completion of treatment(approximately 6 months)
  21 days(3 weeks) for one cycle
C reactive protein | every 3 weeks,up to completion of treatment(approximately 6 months)
  21 days(3 weeks) for one cycle

CONTACTS AND LOCATIONS:
Overall Officials: Wenqi Jiang, MD, Principal Investigator — Department of Medical Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, China State Key Laboratory of Oncology in South China, Sun Yat-Sen University Cancer Center, Guangzhou, China
Locations (1):
- Department of Medical Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wang Y, Wang CQ, Sun P, Liu PP, Yang H, Wang HY, Rao HL, Li S, Jiang WQ, Huang JJ, Li ZM. Phase II Study of Gemcitabine, Peg-Asparaginase, Dexamethasone and Methotrexate Regimen for Newly Diagnosed Extranodal Natural Killer/T-Cell Lymphoma, Nasal Type: Final Analysis With Long-Term Follow-Up and Rational Research for the Combination. Front Oncol. 2022 Jan 24;12:796738. doi: 10.3389/fonc.2022.796738. eCollection 2022. PMID 35141162